CLINICAL TRIAL: NCT07265882
Title: Bed Side Assessment in Patients With Acute Respiratory Failure Under Invasive Mechanical Ventilation
Acronym: BAM
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Pozzi, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: BAM
Record Dates: First submitted 2025-03-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Failure (ARF)
Keywords: respiratory mechanics; ARDS; mechanical ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to learn about the respiratory mechanics in patients undergoing mechanical ventilation. The investigators can achieve this through the offline analysis of data provided by the ventilator. Within the field of respiratory mechanics, the study focuses particularly on the quantification of lung instability.

What does lung instability mean? By this definition, the investigators refer to the part of lung tissue that opens during inspiration and then collapses during the subsequent expiration. The more diseased the lung (for example, in the case of viral pneumonia), the greater the quantity of this tissue.

How is lung instability measured? In the context of the study analysis, lung instability is measured through the analysis of the low flow pressure-volume loop during ventilation. This graph illustrates how the volume of air in the lungs varies in response to the pressures applied by the ventilator during slow inflation and deflation phases. This maneuver is considered quick and safe and has been an integral part of our clinical practice for several years. Through this maneuver, investigators can examine the range of pressures provided by the ventilator during tidal ventilation. To assess lung instability, hysteresis is analyzed, which represents a distinctive characteristic of the pressure-volume loop. Greater hysteresis indicates a higher degree of lung instability.

During the study, investigators will record not only hysteresis but also classical respiratory mechanics parameters (for example, elastance of the respiratory system, i.e., how stiff the lung is), parameters regarding gas exchange (blood oxygen and carbon dioxide levels), biometric data (for example, height and weight), and imaging (CT scans, lung ultrasound, and electrical impedance tomography) to relate them to the degree of lung instability.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing passive mechanical ventilation

Exclusion Criteria:

* hemodynamic instability
* confirmed intracranial hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the reference intensive care unit requiring passive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Statistical prevalence of respiratory system instability , defined as indexed lung hysteresis at PEEP lower than 10 cmH2O. | up to 45 months
  Lung instability is defined as indexed hysteresis > 100. Where:
  * Hysteresis (ml) is calculated as the area enclosed between inspiratory and expiratory limb of the low flow pressure volume loop.
  * indexed hysteresis corresponds to the hysteresis area normalized for the applied driving pressure (plateau pressure minus PEEP)

SECONDARY OUTCOMES:
Description of classical respiratory mechanics related to lung instability | up to 45 months
  Correlate respiratory system compliance (measured as tidal volume divided by driving pressure) with the degree of lung instability (ie indexed hysteresis)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No